CLINICAL TRIAL: NCT03755921
Title: The Effects of Brief and Intensive Therapy for Dysphagia in Patients With Head and Neck Cancer
Brief Title: Brief and Intensive Therapy for Dysphagia in Patients With Head and Neck Cancer
Acronym: dysphagia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Fabrício Edler Macagnan, Clinical professor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TBI2018
Record Dates: First submitted 2018-07-09; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Deglutition Disorders; Dysphagia; Head and Neck Cancer; Radiotherapy; Complications
MeSH Terms: conditions — Deglutition Disorders; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: The control group will receive speech therapy with weekly frequency, and the intervention group will participate in a brief and intensive therapy program that will take place during five days a week for three weeks, totaling fifteen sessions. The sessions will be of 40 minutes and, in both groups, the patients will receive care of individualized form, according to their needs
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief and intensive therapy (Experimental): exercises for swallowing (strength and mobility of oral and pharyngeal muscles) controlling the number of series according to each participant, daily
  Interventions: Other: bried and intensive therapy
- Therapy Weekly (Active Comparator): exercises for swallowing (strength and mobility of oral and pharyngeal muscles) controlling the number of series according to each participant, weekly
  Interventions: Other: bried and intensive therapy

INTERVENTIONS:
Other: bried and intensive therapy — Speech Therapy Exercises

SUMMARY:
According to data in the literature, patients with head and neck cancer, who undergo combined treatment of radio-chemotherapy, have, to a greater or lesser extent, swallowing changes. Most of the time, these patients undergo traditional speech-language interventions, performed weekly. This project proposes a brief and intensive therapy program for dysphagia, with daily interventions, showing that this therapeutic modality generates benefits in a shorter time interval when compared to traditional therapy. This short service period contributes to the reduction of hospital costs and reduces the total number of interventions, which is beneficial for both the patient and the service that performs the care. The present study was to verify the efficacy of a brief and intensive therapy program for dysphagia in patients with head and neck cancer submitted to radio-chemotherapy treatments, since they present, to a greater or lesser extent, changes of swallowing. This is a randomized clinical trial pilot project that will be developed in an oncology hospital. The population of this study is composed of patients diagnosed with head and neck cancer, over 18 years of age, with indication of combined radiotherapy , referred for speech therapy through the Multidisciplinary Oncology Outpatient Clinic of Santa Rita Hospital (AMOHR).

DETAILED DESCRIPTION:
he sample will consist of 20 patients who will be randomized into two groups: 10 in the intervention group with intensive brief therapy and 10 in the control group with traditional weekly therapy. In both groups, instruments related to swallowing assessment and quality of life will be applied before and after speech therapy. The control group will receive speech therapy with weekly frequency, and the intervention group will participate in a brief and intensive therapy program that will take place during five days a week for three weeks, totaling fifteen sessions. The sessions will be of 40 minutes and, in both groups, the patients will receive care of individualized form, according to their needs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients from 18 years of age;
* Diagnosis of head and neck cancer;
* Indication of combined treatment of radio-chemotherapy;

Exclusion Criteria:

* Have performed prior speech and hearing care for at least three months prior to the start of the study;
* Previous history of other neoplasias and / or neurological diseases, according to the participant's report and information of the medical record;
* Cognitive deficits and / or changes in the central nervous system that make it difficult to understand commands (illiterate individuals will have scores of at least 20 points, followed by 25 individuals from 1 to 4 years of study, 26.5 to 5 at 8 years, 28 to 9 to 11 years and finally, 29 to 11 years or more of schooling, according to Brucki et al., 2003).
* Cardiac problems, according to the participant's report and information on the medical chart.
* Do not attend therapy for more than three sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
M. D. Anderson Dysphagia Inventory (MDADI) | 3 months average
  41/5000 quality of life parameter, questionnaire.Questionnaire developed by Chen et al. (2001) and validated by Guedes et al. (2013) With the objective of evaluating the quality of life of patients. consisting of 20 items, involving global, physical, functional and emotional domains, with objective of assessing the impact of dysphagia on the quality of life of patients who underwent treatment of head and neck cancer

SECONDARY OUTCOMES:
Functional Oral Intake Scale | 3 months average
  oral intake, skale. It is composed by a seven-level scale, which graduates oral intake of patients.
  Scale of seven levels, graduates the oral intake of patients. At level 1, the patient is exclusively using an alternative feeding route, with no oral conditions. At levels 2 and 3, it still depends on a consistency. At levels 4,5 and 6 it can be oral total in one of the most consistencies, with or without compensation, but with some restrictions. At level 7, the patient had total oral conditions, without restrictions.
Iowa Oral Performance Instrument (IOPI) | 3 months average
  strength of language, assessment, equipment. Instrument developed in 1992, which allows to evaluate the strength and resistance of the tongue, by inserting a bulb into the oral cavity. The patient should lift the dorsum, and / or the anterior portion of the tongue against this bulb, pushing as hard as he can. Afterwards, the pressure transducer circuits of the apparatus will detect bulb compression, indicating the peak pressure result (Solomon et al, 2008; Robins et al, 2007).
Deglutition evaluation | 3 months average
  evaluation of swallowing, protocol. In the structural evaluation (normal or altered), morphological (normal or altered) deglutitionstrength (normal or flaccid), mobility (normal or reduced), coordination (normal or altered) and sensitivity (normal or reduced), swallowing reflex (present or ausent), clinical signs suggestive of penetration / aspiration (present or ausent).

IPD SHARING:
Plan to Share IPD: No